CLINICAL TRIAL: NCT05745402
Title: A Longitudinal Study of the Effectiveness of the Mobility Checkup for Older Adults: Feasibility in the 'Year 1' Cohort
Brief Title: Longitudinal Study to Determine the Effectiveness of the Mobility Checkup for Older Adults
Acronym: LEMCOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: College of St. Scholastica, Inc. (Other)
Responsible Party: Principal Investigator, Alexandra Borstad, Associate Professor, College of St. Scholastica, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1234
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobility Checkup Intervention (Experimental): 45-minute Mobility checkup that includes 5 physical performance measures and education based on outcomes compared to age and gender normative values.
  Interventions: Behavioral: Mobility Checkup for older adults

INTERVENTIONS:
Behavioral: Mobility Checkup for older adults — The Mobility Checkup (MC) for older adults is a 45-minute preventative physical therapy visit designed to maintain mobility during aging. It has two parts, measurement (25 minutes) and education (20 minutes). The 5 standardized measures of physical performance in the MC are Walking speed, single leg stance time (balance), Five rep sit to stand (muscular endurance, transitions), 6-meter walk test (general endurance), and Timed up from floor test (transitions). Participants are provided education structured into 4 elements. 1. They are told their performance scores 2. They are shown how their performance scores on each of the measures compare to age and sex-referenced normative values 3. They are provided information about what their performance predicts about their health 4. They are referred to an appropriate provider if there was a health or safety concern during their MC or they are educated to follow the recommendations for physical activity that are recommended by the CDC.

SUMMARY:
The investigators are developing a new, preventative physical therapy model of care for older adults called Mobility Checkup (MC). Proposed as an annual visit, the MC includes measurement of physical performance and education regarding the importance of maintaining mobility for overall health. The purpose of this study is to determine the feasibility of and begin data collection for, a longitudinal study of the effectiveness of the Mobility Checkup with a small cohort. This activity will evaluate the feasibility of recruitment and implementation of this longitudinal effectiveness study.

DETAILED DESCRIPTION:
Healthy aging is defined as "the process of developing and maintaining the functional ability that enables well-being in older age" and includes mobility. Mobility disability (i.e., the inability to walk 400 meters and climb a flight of stairs without assistance) is the most prevalent form of disability for older adults in the United States. Unlike blood pressure or body mass index, physical performance measures such as walking speed help identify and predict preclinical mobility disability, but are rarely used in routine medical care. This is a missed opportunity, particularly for older adults, who may experience a subtle decline in physical performance that leads to mobility disability.

The position of the American Physical Therapy Association is that all people should have an annual physical therapy visit to optimize movement and promote health, wellness, and fitness; and slow the progression of impairments of body functions and structures, activity limitations, and participation restrictions.

Recommendations support preventive care for maintaining mobility. However, a model of care specific to preventing mobility disability in older adults is not common practice. Evidence suggests routine screening can predict mobility disability in older adults and that activity-based interventions prevent it.

The is year 1 of a longitudinal study that will determine the feasibility of an effectiveness study of a Mobility Checkup, an annual preventive visit within a model of physical therapy care. The Mobility Checkup prioratizes educating older adults on the value of physical performance as an indicator of health and aims to maintain mobility and reduce mobility disability among participants. Ultimately, this new model of care could result in a cost-effective tool to establish baseline physical performance and identify and prevent preclinical and mobility disabilities in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Walk independently with or without an assistive device

Exclusion Criteria:

* Experiencing short-term condition affecting their mobility
* Cardiac procedure or myocardial infarction (heart attack) in the last 6 months
* Has a guardian who is responsible for their healthcare decisions

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
LASA Physical Activity Questionnaire (LAPAQ) | one year
  Questionnaire designed to measure the amount of physical activity a person completed over the last two weeks.

SECONDARY OUTCOMES:
The 6-minute walk test | one year
  In the 6-minute walk test the distance in meters a person can walk in 6 minutes is measured as evidence of their endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- College of St. Scholastica-Health Science Center, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lieberz D, Borgeson H, Dobson S, Ewings L, Johnson K, Klaysmat K, Schultz A, Tasson R, Borstad AL. A Physical Therapy Mobility Checkup for Older Adults: Feasibility and Participant Preferences From a Discrete Choice Experiment. J Patient Cent Res Rev. 2022 Jan 17;9(1):24-34. doi: 10.17294/2330-0698.1874. eCollection 2022 Winter. PMID 35111880